CLINICAL TRIAL: NCT06782880
Title: Efficacy and Safety of Fecal Microbiota Transplantation for the Prevention of Early-onset Infectious Complications After Orthotopic Liver Transplantation
Brief Title: Fecal Microbiota Transplantation for the Prevention of Infectious Complications After Liver Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMT-OLT; Bando RF-2021-12373311 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-12-03; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-11

CONDITIONS: Fecal Microbiota Transplantation; Orthotopic Liver Transplantation; Multi-drug Resistant Bacteria
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: All adult patients listed or being evaluated for enlistment for OLT for various etiologies are eligible for inclusion in the present study. Study enrollment will start after the favorable opinion of the Ethics Committee and the authorization by the General Manager of IRCCS AOUBO, in May 2023, indicatively, and will last 24 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heterologous FMT (Experimental): Heterologous feces will be processed from routinely screened universal donors. Adult patients listed or being evaluated for enlistment for OLT for various etiologies are eligible for Fecal Microbiota Transplantation. Fecal material must be infused by enema or colonoscopy.
  Interventions: Procedure: Fecal microbiota transplantation (FMT)
- Homologous FMT (Placebo Comparator): The control arm will undergo autologous FMT after enrollment. Autologous feces will be collected by each patient the day before each FMT in both study arms. This will guarantee adequate patients' stool collection in order to subsequently store the fecal samples for autologous FMT and ensure blinding.
  Interventions: Procedure: Fecal microbiota transplantation (FMT)

INTERVENTIONS:
Procedure: Fecal microbiota transplantation (FMT) — To assess if heterologous FMT is more effective than autologous FMT in reducing the rate of major infection episodes within 6-months after OLT.

SUMMARY:
The increasing emergence and spread of MDRB represents a major public health problem, with higher mortality in patients experiencing infections. Cirrhotic patients listed for OLT and after OLT are at high risk of MDRB colonization or infection due to the large use of broad-spectrum antibiotics in the post-transplant setting. Therefore, effective decolonization strategies in this particular setting are urgently needed. The investigators hypothesize that heterologous FMT can reduce infections rates in the pre-and post- OLT setting by MDRB decolonization and restoration of a more physiological microbiome.

DETAILED DESCRIPTION:
The study is a double-blind, single-center, randomized controlled trial and will be offered consecutively to every adult patient on the liver transplant list.

Enrolled patients will be randomized (1:1) and assigned to either the heterologous or autologous fecal microbiota transplantation.

The intervention of the trial is heterologous fecal microbiota transplantation, which involves the administration of fecal material from a healthy donor into the intestine of the enrolled patient. Fecal samples will be collected every three months and before each microbiota transplant for evaluation of fecal microbiota composition. Gut permeability tests will be evaluated at enrollment and after the first fecal transplantation. Moreover, clinical and microbiota assessments will be performed after liver transplantation. All other planned assessments are part of the normal course of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age≥18 years) patients listed for OLT for various etiologies.
* Patient's consent to participate in the study

Exclusion Criteria:

* Previous total colectomy
* Pregnancy or breastfeeding
* Patients on oral or intravenous antimicrobial agents
* HIV positive and not well controlled on antiretroviral therapy, or CD4+ <200/ mm3
* Active SARS-CoV-2 infection
* Neutropenia <0.5X10^9/L
* Toxic megacolon
* Contraindications to colonoscopy
* Any conditions for which, according to the physician, FMT endangers the patient's health
* History of hypersensitivity to macrogol contained in bowel preparations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
To assess if heterologous FMT is more effective than autologous FMT in reducing the rate of major infection episodes within 6-months after OLT. | At 6 months after OLT
  Incidence of clinically severe infections (sepsis, severe sepsis, septic shock)

SECONDARY OUTCOMES:
Incidence of adverse events after FMT | 3 years
  To evaluate the safety profile of both heterologous and autologous FMT in patients enlisted for OLT and the relationship between fecal microbiota composition and the gastrointestinal permeability profile before and after FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbara, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No